CLINICAL TRIAL: NCT06349681
Title: Describe Relationship Between qCON and qNOX of the CONOX Monitor During General Anesthesia Perfromed With Propofol and Remifentanil Target Controlled Infusion (TCI)
Brief Title: Describe Relations Between qCON and qNOX Indicies During Propofol-Remifentanil General Anesthesia
Status: Recruiting | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Federico Linassi, Principal Investigator, University of Padova
Other Study IDs: CONOXBird
Record Dates: First submitted 2024-03-24; First posted 2024-04-05 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia Brain Monitoring
Keywords: Anesthesia brain Monitoring; TIVA-TCI; CONOX

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CONOX is a neuromonitoring EEG- device for sedation (qCON) and analgesia (qNOX) monitoring during general anesthesia.

It is unknown on how the indicies can differentiate themselves so aim of this study is to determine the relationship bewtween the 2 indicies.

DETAILED DESCRIPTION:
CONOX is a neuromonitoring EEG- device for sedation (qCON) and analgesia (qNOX) monitoring during general anesthesia.

It is unknown on how the indicies can differentiate themselves so aim of this study is to determine the relationship bwtween the 2 indicies, as well as with EMG, Concentration of Propofol (CeP) and Remifentanil (CeR) during Total Intravenous Anesthesia with Target Controlled Infusion (TIVA-TCI).

ELIGIBILITY:
Inclusion Criteria:

* Undergo general anaesthesia with Targeted Controlled Infusion of Propofol (Eleveld or Schnider model) and Remifentanil (Minto model) and CONOX monitoring

Exclusion Criteria:

* Neurological disease
* Psychiatric disease
* Obesity
* Locoregional anesthesia

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing brast cancer surgery with general anesthesia with Propofol and Remifentanil TCI will be recruited
Sampling Method: Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between qCON and qNOX | CONOX values will be recorded from start of anesthesia to the return of responsiveness at the end of surgery
  qCON and qNOX values from CONOX monitor will be compared

SECONDARY OUTCOMES:
Correlation between qCON and concentrations of Propofol(CeP) | CONOX and TCI values will be recorded from start of anesthesia to the return of responsiveness at the end of surgery
  qCON and CeP values from CONOX monitor and infusion pump will be compared
Correlation between qNOX and concentrations of Remifentanil (CeR) | CONOX and TCI values will be recorded from start of anesthesia to the return of responsiveness at the end of surgery
  qNOX and CeR values from CONOX monitor and infusion pump will be compared

CONTACTS AND LOCATIONS:
Locations (1):
- Treviso Regional Hospital, Treviso, TV, Italy

IPD SHARING:
Plan to Share IPD: Undecided